CLINICAL TRIAL: NCT03388918
Title: Future Patient - Telerehabilitation of Heart Failure Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University (Other)
Collaborators: Aage og Johanne Louis-Hansens Fond (Other); Viewcare A/S (Unknown); Laboratory of Welfare Technologies - Telehealth & Telerehabilitation, SMI, Department of Health Science and Technology, Aalborg University (Unknown); Regionshospitalet Viborg, Skive (Other); Technical University of Denmark (Other); University of Aarhus (Other); Danish Heart Foundation (Other); Viborg Healthcare Center (Unknown); Skive Healthcare Center (Unknown); Odense University Hospital (Other); Department of Computer Science, AAU (Unknown)
Responsible Party: Principal Investigator, Birthe Dinesen, Professor, Aalborg University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: N-20160055
Record Dates: First submitted 2017-08-24; First posted 2018-01-03 (Actual); Last update posted 2021-05-27 (Actual); Status verified 2021-05

CONDITIONS: Heart Failure NYHA Class I; Heart Failure NYHA Class II; Heart Failure NYHA Class III; Heart Failure NYHA Class IV; Acute Decompensated Heart Failure
Keywords: Quality of life; Telerehabilitation; Cardiac patients; Heart failure
MeSH Terms: conditions — Heart Failure | interventions — Telerehabilitation

STUDY DESIGN:
Intervention Model Description: Randomised controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The intervention group has three steps:
  Step I: Titration of medicine ( 0-3 months)
  Step II: Telerehabilitation program at healthcare center or by call center ( 3 months)
  Step III: Rehabilitation in everyday life ( 6 months)
  The patients is monitoring vital signs such as blood pressure, pulse, weight, steps, respiration, and sleep. Have access to a Heart Portal that is an information cite on heart failure. Via the portal patients can see measured values & communicate with staff. Every other week the patients fill in an online questionnaires on symptoms, sleep and well being.
  Interventions: Device: Telerehabilitation
- Traditional rehabilitation group (No Intervention): This group follows the International Cardiac Guidelines. There are three steps in this arm:
  Step I: Titration of medicine (3 months).
  Step II: Traditional rehabilitation at the healthcare center ( 3 months).
  Step III: Everyday life with HF ( 6 months)
  The participants do not have access to the Heart Portal and is not monitoring any vital signs.

INTERVENTIONS:
Device: Telerehabilitation — Blood pressure (A&D Medical UA 767PBT), weight (A&D Medical UC-321PBT), step counters(Fitbit Zip & Charge), sleep sensor (Beddit 3), tablet (iPAD Air 2) & transmitter (Qualcomm Life, QWH-HUB-V1.0E)
  Arms: Intervention group

SUMMARY:
The idea behind the Future Patient research project is to develop a telerehabilitation program and tools for patients with heart failure.

The hypothesis for this study is that participation in a telerehabilitation program for patients with heart failure will increase the patients' quality of life and multi-parametric (subjective and objective) individualized monitoring in a telerehabilitation program for patients with heart failure will increase detection of worsening of symptoms and avoid future hospitalization of the HF-patients.

DETAILED DESCRIPTION:
The overall aim is to test, implement and evaluate a telerehabilitation program for patients with heart failure from clinical, psychosocial, health literacy and e-health literacy, inter-organizational, health economic and technical perspectives.

Furthermore, this study has sub aims:

* To increase the quality of life for patients with Heart Failure (HF)
* To optimize the medical treatment of patients with HF
* To perform multi-parametric (subjective and objective) individualized monitoring in order to detect worsening of symptoms and avoid hospitalizations
* To increase physical activities for patients with heart failure in everyday life in a telerehabilitation program
* To facilitate patient-initiated self-care management actions upon the following early detection of changes in source data (steps taken, weight, blood pressure, pulse, sleep, illness perception, motivation, anxiety and depression)
* To evaluate patients health literacy and e-health literacy participating in a telerehabilitation program and rehabilitation program
* To test and evaluate the Heart Portal - a digital toolbox for improved self-management for patients with heart failure and their relatives
* To explore the experiences and perspectives of the patients and their relatives when being part of a telerehabilitation program
* To test and evaluate a cross sector communication platform from a patient and healthcare professional perspective
* To perform a cost-effectiveness analysis of total costs of healthcare and rehabilitation services

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with HF according to New York Heart Association (NYHA) Class I-IV with max 20 % in class I or who have a current hospitalization for acute decompensated HF within the past two weeks
* Adults (18 years or older); no upper age limit
* Patients living in Viborg and Skive Municipality
* Living at home and capable of caring for him/herself
* Have basic computer skills or a relative who have basic computer skills
* Informed consent to participate in a telerehabilitation program
* May have a pacemaker

Exclusion Criteria:

* Pregnancy
* Drug addiction defined as the use of cannabis, opioids or other drugs
* Previous neurologic, musculoskeletal or cognitive disability or active psychiatric history (as noted in the medical record) other than depression or anxiety related to cardiac or other chronic illness
* Lack of ability to cooperate
* Does not speak Danish

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2016-12-21 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2019-08-01 (Actual)

PRIMARY OUTCOMES:
Increased quality of life | Intervention group: At baseline, week 2,4,6,8,10,12,14,16,18,20,22,24,26,28,30,32, 34,36,38,40,42,44,46,48,50,52 Control group: Baseline, 6 & 12 months
  Increased quality of life as measured by a moderate change (10 points) in quality of life measured by Kansas City Questionnaire (KCCQ)

SECONDARY OUTCOMES:
Time from baseline to optimized medical treatment | For both intervention and control group: From date of randomization until the date of first documented progression with medical treatment, assessed up to 4 months
  Time for optimizing medicine
All cause hospitalization | For both intervention and control group: 6 months
  All-cause hospitalization at end of rehabilitation
Steps taken | Intervention group: Everyday for 12 months
  Numbers of steps taken in the intervention group
Development of bloodpressure | Intervention group: Blood pressure (mmHG) from date of randomization twice a week assessed up to 3 months
  Intervention group: Blood pressure (mmHG)
Development of pulse | Intervention group: Pulse from date of randomization and every day in 12 months
  Intervention group: Pulse ( numbers per minutes)
Development of weight | Intervention group: Weight from date of randomization and every day in 12 months
  Intervention group: Weight (Kilograms)
Sleep | Intervention group: Sleep from date of randomization and accessed up to 12 months
  Intervention group: Sleep ( numbers of hours per night)
Illness perception | For Intervention and control group: At baseline, 6 & 12 months
  Positive changes in illness perceptions, from dysfunctional to functional measured by Illness perception questionaire
Motivation | For both intervention and control group: At baseline, 6 & 12 months
  Changes from extrinsic to intrinsic motivation measured from baseline to end of rehabilitation and 6 months after end of rehabilitation measured by Health Climate Change Questionaire
Anxiety and depression | For both intervention and control group: At baseline, 6 & 12 months
  Explore whether levels of anxiety and depression in the intervention group are lower or equivalent to the control group measured by Hospital Anxiety and Depression Scale (HADS) questionnaire
Health- literacy | For both intervention and control group: At baseline
  Health literacy in intervention and control group measured by Health Literacy Questionnaire (Danish validated version HLQ) by units on a scale
eHealth literacy | For both intervention and control group: At baseline, 6 & 12 months
  Improvement in e-health literacy in intervention and control group measured by eHealth Literacy Questionnaire (Danish validated version eHLQ) by units on a scale
Experiences of using the Heart portal | For intervention group: 6 & 12 months
  Qualitative exploration of experiences of HF patients, relatives and healthcare professionals use of the Heart portal
Costs of healthcare and rehabilitation services | For both intervention and control group: 6 months
  Number of hospitalizations, number of contacts with heart failure clinic, days at hospital, contacts with general practitioners, number of participations in rehabilitation activities at healthcare center between intervention and control group

CONTACTS AND LOCATIONS:
Overall Officials: Birthe Dinesen, PhD, Principal Investigator — Aalborg University; Malene Hollingdal, MD, PhD, Study Director — Central Jutland Regional Hospital; Jens Refsgaard, MD, PhD, Study Director — Central Jutland Regional Hospital
Locations (1):
- Cardiology Ward, Viborg Hospital, Viborg, Denmark

IPD SHARING:
Plan to Share IPD: No
No plan for sharing protocol as we are applying for patent.

REFERENCES:
- [Derived] Spindler H, Dyrvig AK, Schacksen CS, Anthonimuthu D, Frost L, Gade JD, Kronborg SH, Mahboubi K, Refsgaard J, Dinesen B, Hollingdal M, Kayser L. Increased motivation for and use of digital services in heart failure patients participating in a telerehabilitation program: a randomized controlled trial. Mhealth. 2022 Jul 20;8:25. doi: 10.21037/mhealth-21-56. eCollection 2022. PMID 35928510
- [Derived] Skov Schacksen C, Dyrvig AK, Henneberg NC, Dam Gade J, Spindler H, Refsgaard J, Hollingdal M, Dittman L, Dremstrup K, Dinesen B. Patient-Reported Outcomes From Patients With Heart Failure Participating in the Future Patient Telerehabilitation Program: Data From the Intervention Arm of a Randomized Controlled Trial. JMIR Cardio. 2021 Jul 2;5(2):e26544. doi: 10.2196/26544. PMID 34255642
- [Derived] Dinesen B, Dittmann L, Gade JD, Jorgensen CK, Hollingdal M, Leth S, Melholt C, Spindler H, Refsgaard J. "Future Patient" Telerehabilitation for Patients With Heart Failure: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2019 Sep 19;8(9):e14517. doi: 10.2196/14517. PMID 31538944